CLINICAL TRIAL: NCT00005072
Title: Phase I/II Study Evaluating the Safety and Efficacy of Leuvectin Immunotherapy for the Treatment of Locally Recurrent Prostate Cancer Following Radiation Therapy (Summary Last Updated: 02/2001)
Brief Title: Leuvectin in Treating Patients With Locally Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development in prostate cancer indication halted
Sponsor: Vical (Industry)
Collaborators: Jonsson Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCL-1102-203; UCLA-9906108 (Other: UCLA); CDR0000067677 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1721 (Other: NCI)
Record Dates: First submitted 2000-04-06; First posted 2003-11-04 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuvectin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leuvectin (Experimental): Leuvectin
  Interventions: Biological: Leuvectin

INTERVENTIONS:
Biological: Leuvectin — 1000 ug of Leuvectin injected intratumorally
  Other Names: Interleukin-2 (IL-2) plasmid DNA/lipid complex

SUMMARY:
RATIONALE: Inserting the gene for interleukin-2 into a person's prostate cancer cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of Leuvectin in treating patients who have locally recurrent prostate cancer after receiving treatment with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and tolerability of Leuvectin in patients with locally recurrent organ-confined prostate cancer after radiotherapy. II. Determine the efficacy of this regimen in preventing or delaying manifestations of disease progression as demonstrated by biochemical failure or clinical recurrence in this patient population.

OUTLINE: This is an open-label, multicenter study. Patients receive Leuvectin intraprostatically over 10-30 seconds under transrectal ultrasound guidance on days 0 and 14. Patients are re-evaluated at week 10. Treatment repeats every 10-11 weeks or 1-6 days after completion of each week 10 re-evaluation for a maximum of 3 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 1 year and then every 6 months for 2 years in the absence of disease progression.

ACTUAL ACCRUAL: A total of 25 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally recurrent organ-confined prostate cancer after external beam radiotherapy, radiation seed implants, or cryosurgery. Gleason score of at least 6. Prostate specific antigen values (PSA) of at least 1.0 ng/mL with 2 consecutive rises in PSA at least 2 weeks apart, of which the second increase is greater than the first, after achieving a nadir. Must have at least 3 recorded PSA values over a minimum of the last 3 months to determine the slope. Patients must have declined additional conventional treatment or be ineligible for conventional treatment of their prostate cancer. No metastasis by bone scan. No significant central nervous system (CNS) disease.

PATIENT CHARACTERISTICS: Age: 18 and over. Performance status: Karnofsky 80-100% OR Eastern Cooperative Oncology Group (ECOG) 0 or 1. Life expectancy: Not specified. Hematopoietic: White blood cell count (WBC) greater than 3,000/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 9.0 g/dL. Hepatic: Bilirubin normal. Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) less than 3 times upper limit of normal. Albumin greater than 3 g/dL. Prothrombin time (PT) and partial thromboplastin time (PTT) normal. Hepatitis B surface antigen negative. Renal: Creatinine normal. Cardiovascular: No uncontrolled hypertension. No significant cardiovascular disease, e.g.: History of ventricular dysfunction; Congestive heart failure; Symptoms of coronary artery disease; History of any ventricular arrhythmia; Prior myocardial infarction. Other: HIV negative. Fertile patients must use effective double-barrier contraception during and for 3 months after study participation. No active autoimmune disease. No active infection requiring IV antibiotics. No uncontrolled diabetes mellitus. No significant psychiatric disorder that would preclude study. No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer.

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior Leuvectin. Chemotherapy: At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or hydroxyurea). Endocrine therapy: No prior hormonal therapy for prostate cancer. Radiotherapy: See Disease Characteristics. At least 3 weeks since prior radiotherapy. Surgery: At least 1 month since prior intrathoracic or intra-abdominal surgery. At least 2 weeks since other prior major surgery. Other: At least 10 days since prior anticoagulants or non-steroidal anti-inflammatory agents. No neoadjuvant or other concurrent anticancer drug therapy. No concurrent immunosuppressive drugs. No other concurrent experimental therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2000-11; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Safety of Leuvectin

CONTACTS AND LOCATIONS:
Overall Officials: Arie Belldegrun, MD, FACS, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio